CLINICAL TRIAL: NCT00016250
Title: A Randomized Phase II Study of Two Shcedules of Ro 31-7453 in Patients With Metastatic (Dukes' D) Colorectal Carcinoma (CRC) Who Have Failed Both Fluoropyrimidine and Irinotecan Chemotherapy
Brief Title: Ro 31-7453 in Treating Patients With Recurrent or Refractory Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 00-139; CDR0000068613 (Registry Identifier: PDQ (Physician Data Query)); ROCHE-16113; ROCHE-RO31-7453; NCI-G01-1945
Record Dates: First submitted 2001-05-06; First posted 2003-10-15 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

INTERVENTIONS:
Drug: MKC-1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase II trial to compare the effectiveness of two different regimens of Ro 31-7453 in treating patients who have recurrent or refractory metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the objective disease rate of patients with recurrent or refractory metastatic colorectal cancer treated with two dose schedules of Ro 31-7453.
* Compare the safety and tolerability of these regimens in these patients.
* Compare the response duration in patients treated with these regimens.
* Compare the time to progression and time to treatment failure in patients treated with these regimens.
* Determine the pharmacokinetic profiles of Ro 31-7453 and its major metabolites in these patients.
* Compare the overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, open label, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral Ro 31-7453 twice daily on days 1-4. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral Ro 31-7453 twice daily on days 1-14. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 28 days and then every 3 months.

PROJECTED ACCRUAL: Approximately 160 patients (49 per treatment arm plus 61 additional patients in the arm determined to be most effective) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the colon or rectum
* Bidimensionally measurable disease

  * At least 2.0 x 2.0 cm
* Failed prior fluoropyrimidine and irinotecan chemotherapy in adjuvant or metastatic setting

  * Must have had disease progression while receiving chemotherapy OR
  * If received fluorouracil with or without irinotecan in adjuvant setting, must also have failed therapy with these agents in metastatic setting (unless manifesting metastatic disease during adjuvant therapy)
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 9 g/dL
* Absolute neutrophil count at least 1,500/mm^3
* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 2.5 ULN (5 times ULN if bone or liver metastases present)

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No New York Heart Association class III or IV congestive heart failure
* No myocardial infarction within the past 6 months

Gastrointestinal:

* No bowel obstruction
* No active uncontrolled malabsorption syndrome

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No other prior malignancy within the past 5 years except carcinoma in situ of the cervix or non-melanoma skin cancer
* No other active cancers, including stable disease on adjuvant therapy
* No other medical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Chemotherapy
* At least 2 weeks since prior biologic therapy and recovered

Chemotherapy:

* See Disease Characteristics
* No more than 2 prior cytotoxic chemotherapy regimens for metastatic disease
* Monoclonal antibody (MOAB) therapy and antiangiogenic agents not included as prior cytotoxic chemotherapy
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* No prior total gastrectomy

Other:

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States